CLINICAL TRIAL: NCT05004480
Title: Influence of Surgical Mask on Functional Capacity and Quality of Life During Controlled Endurance Exercise in Sedentary Adults
Brief Title: Influence of Mask on Functional Capacity and Quality of Life During Controlled Endurance Exercise in Sedentary Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Elbanna, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Personal
Record Dates: First submitted 2021-07-27; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Sedentary Adults
Keywords: Surgical mask; Functional capacity; Quality of life; Aerobic exercise
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Subjects had randomly divided into two groups. All will do aerobic exercise in form of treadmill but Group (A) will do while wearing surgical mask and Group (B) without surgical mask. To detect the Influence of surgical mask on functional capacity and quality of life during controlled endurance exercise in sedentary adults
Who Masked: Participant
Masking Description: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Mask Group (Experimental): participants of both sexes who will perform controlled endurance exercise on treadmill while wearing surgical mask
  Interventions: Device: Treadmill
- Non mask Group (Experimental): participants of both sexes who will perform controlled endurance exercise on treadmill without wearing surgical mask
  Interventions: Device: Treadmill

INTERVENTIONS:
Device: Treadmill — Electronic treadmill, Hammer T-2000 Treadmill, 2,5 HP - 140 Kilograms

SUMMARY:
Subjects had randomly divided into two groups. All will do aerobic exercise in form of treadmill but Group (A) will do while wearing surgical mask and Group (B) without surgical mask. To detect the Influence of surgical mask on functional capacity and quality of life during controlled endurance exercise in sedentary adults

DETAILED DESCRIPTION:
Group (A):

1. Each subject will sign a consent form after receiving a detailed explanation about the procedure.
2. Functional capacity and Quality of life will be evaluated before the start of the training.
3. Subjects in group A will wear surgical mask before starting of the session. 4.3 sessions will be done every week for 3 months.

5.The session will start with warming up for 5 minutes then 25 minutes of aerobic exercise on the treadmill with moderate intensity followed by cooling down for 5 minutes.

6.After finishing the program, the participant will be evaluated to detect the effect of the exercise.

Group (B):

1. Each subject will sign a consent form after receiving a detailed explanation about the procedure.
2. Functional capacity and Quality of life will be evaluated before the start of the training.
3. Subjects in group A will not wear any mask during the session. 4.3 sessions will be done every week for 3 months.

5.The session will start with warming up for 5 minutes then 25 minutes of aerobic exercise on the treadmill with moderate intensity followed by cooling down for 5 minutes.

6.After finishing the program, the participant will be evaluated to detect the effect of the exercise.

ELIGIBILITY:
Inclusion Criteria:

* 100 participants
* 30 to 40 years of age
* both sex

Exclusion Criteria:

* uncontrolled cardiopulmonary conditions,
* sever un treated orthopedic condition
* uncontrolled neurological conditions,)
* uncontrolled diabetes,
* claustrophobia,
* pregnancy
* Recent COVID-19 infection,)

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-10-20 (Estimated)

PRIMARY OUTCOMES:
Influence of surgical mask on Blood pressure during controlled endurance exercise in sedentary adults | three months
  Measuring Blood pressure before and after the all program
Influence of surgical mask on Resting and post exercise heart rate during controlled endurance exercise in sedentary adults | three months
  Measuring Resting and post exercise heart rate before and after the all program
Influence of surgical mask on resting and post exercise respiratory rate during controlled endurance exercise in sedentary adults | three months
  Measuring resting and post exercise respiratory rate before and after the all program
Influence of surgical mask on oxygen saturation, maximum oxygen consumption during controlled endurance exercise in sedentary adults | three months
  Measuring oxygen saturation, maximum oxygen consumption before and after the all program
Influence of surgical mask on quality of life during controlled endurance exercise in sedentary adults | three months
  quality of life will be measured using short form quality of life 36 questionnaire, with score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.

SECONDARY OUTCOMES:
Influence of surgical mask on rate of perceived exertion during controlled endurance exercise in sedentary adults | three months
  rate of perceived exertion will be measured by Borg scale with score ranged from 6-20 before and after intervention.
Influence of surgical mask on submaximal exercise capacity during controlled endurance | three months
  submaximal exercise capacity will be detected by six-minutes walking test and the distance which will be obtained will be measured by meter before and after the all program

CONTACTS AND LOCATIONS:
Overall Officials: Rana H El Banna, PHD, Principal Investigator — Outpatient clinic faculty of physical therapy at Cairo University
Locations (1):
- Outpatient clinic faculty of physical therapy at Cairo University, Giza, Egypt